CLINICAL TRIAL: NCT00878449
Title: A Phase 1 Study Evaluating the Safety of ABT-263 in Combination With Etoposide/Cisplatin in Subjects With Cancer
Brief Title: A Study Evaluating the Safety of ABT-263 in Combination With Etoposide/Cisplatin in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-234
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — navitoclax; PE regimen

ARMS (1):
- ABT-263 + etoposide/cisplatin (Experimental)
  Interventions: Drug: ABT-263; Drug: etoposide/cisplatin

INTERVENTIONS:
Drug: ABT-263 — 150mg of ABT-263 is taken daily for 3 out of 21 days. This is a dose escalation study, therefore the dose of ABT-263 will change throughout the study.
Drug: etoposide/cisplatin — etoposide = 100 mg/m2 Days 1-3 of each Cycle; Max duration 6 cycles. cisplatin = 75 mg/m2 Day 1 of each Cycle; Max duration 6 cycles

SUMMARY:
This is a Phase 1 Study Evaluating the Safety of ABT-263 in Combination with Etoposide/Cisplatin in Subjects with Small Cell Lung Cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Must be greater then or equal to18 years of age;
* For dose escalation subject must have histologically and/or cytologically documented cancer for which etoposide/cisplatin has been determined to be an appropriate therapy. For expanded safety cohort subject must have histologically and/or cytologically documented SCLC for which etoposide/cisplatin has been determined an appropriate therapy;
* Subject has an ECOG performance score of less then or equal to 1; Evaluable and/or measurable disease by CT or MRI per RECIST criteria;
* Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the 1st dose of study drug;
* Must have adequate renal and hepatic function, per local laboratory reference range at Screening as follows:

  * ANC greater then or equal to 1500/mcL,
  * Platelets greater then or equal to 150,000/mm^3,
  * Hemoglobin greater then or equal to 10.0 g/dL,
  * Serum creatinine less then or equal to 1.5 mg/dL or calculated creatinine clearance greater then or equal to 50 mL/min; Na greater then 130 mmol/L,
  * Alkaline Phosphatase, AST and ALTless then or equal to 2.5 x ULN ;Bilirubin less then or equal to 1.5 x ULN.Subjects with liver mets may have ALP, AST and ALT less then or equal to 5.0 x ULN, Subjects with bone mets may have Alkaline Phosphatase less then or equal to 5.0 x ULN,
  * Subjects with Gilbert's Syndrome may have a Bilirubin greater then 1.5 x ULN,
  * Coagulation: aPTT, PT, less then or equal to 1.2 x ULN;
* Life expectancy of at least 30 days;
* Female subjects must be surgically sterile, postmenopausal (for at least 1 year), or have negative results for a pregnancy test;
* Female subjects not surgically sterile or postmenopausal (for at least one year) and non-vasectomized male subjects must practice at least one method of birth control.

Exclusion Criteria:

* Subject exhibits evidence of other uncontrolled condition(s) including, but not limited to: active systemic infection, diagnosis of fever or neutropenia within 1 week of 1st dose;
* Subject has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding;
* Subject is currently receiving or requires anticoagulation therapy;
* Subject has active immune thrombocytopenic purpura, autoimmune hemolytic anemia or a history of being refractory to platelet transfusions (within 1 year prior to 1st dose of study drug);
* Subject has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis;
* Subject has a significant history of CV disease, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease;
* Female subject is pregnant or breast-feeding;
* Subject has tested positive for HIV;
* Subject has a history of other active malignancies within 3 years prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin, previous malignancy confined and surgically resected with curative intent;
* Subject has received any anti-cancer therapy within 14 days prior to 1st dose of study drug;
* Subject has received steroid therapy for anti-neoplastic intent within 7 days prior to 1st dose of study drug;
* Subject has received aspirin within 7 days prior to 1st dose of study drug;
* Subject has received radio-immunotherapy within 6 months prior to 1st dose of study drug; Subject has received an antibody therapy or other biologics (with the exception of colony stimulating factors [G-CSF,GM-CSF] or erythropoietin) within 28 days prior to 1st dose of study drug;
* Subject has a hypersensitivity to platinum-containing compounds or etoposide;
* Subject has consumed grapefruit within 3 days prior to 1st dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of ABT-263 when administered in combination with etoposide/cisplatin in subjects with Cancer. | Weekly
Characterize the pharmacokinetics of ABT-263 when administered in combination with etoposide/cisplatin . | Weekly
Determine the maximum tolerable dose (MTD) of ABT-263 when administered in combination with etoposide/cisplatin. | Weekly
Determine the recommended Phase 2 dose (RPTD) of ABT-263 when administered in combination with etoposide/cisplatin. | Weekly

SECONDARY OUTCOMES:
Evaluate preliminary data regarding progression free survival (PFS). | Bi-monthly
Evaluate preliminary data regarding objective response rate (ORR). | Bi-monthly
Evaluate preliminary data regarding time to tumor progression (TTP). | Bi-monthly
Evaluate preliminary data regarding overall survival (OS). | Bi-monthly
Evaluate preliminary data regarding duration of overall response. | Bi-monthly
Evaluate preliminary data regarding Eastern Cooperative Oncology Group (ECOG) performance status. | Bi-monthly
Evaluate biomarkers | Bi-monthly
  Define the relationship between disease state (related to patient selection and monitoring), B-Cell Lymphoma 2 (Bcl-2) family protein expression, and potential response to the proposed therapy ABT-263 and etoposide/cisplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — AbbVie
Locations (7):
- United States (7):
  - Site Reference ID/Investigator# 13323, Chicago, Illinois
  - Site Reference ID/Investigator# 12841, Maywood, Illinois
  - Site Reference ID/Investigator# 12303, Baltimore, Maryland
  - Site Reference ID/Investigator# 12305, Boston, Massachusetts
  - Site Reference ID/Investigator# 20381, Boston, Massachusetts
  - Site Reference ID/Investigator# 43505, Detroit, Michigan
  - Site Reference ID/Investigator# 13322, New Brunswick, New Jersey

REFERENCES:
- [Background] Pietanza MC, Rudin CM. Novel therapeutic approaches for small cell lung cancer: the future has arrived. Curr Probl Cancer. 2012 May-Jun;36(3):156-73. doi: 10.1016/j.currproblcancer.2012.03.005. Epub 2012 Apr 10. No abstract available. PMID 22495056